CLINICAL TRIAL: NCT03107871
Title: Randomized Controlled Trial of Valganciclovir for Cytomegalovirus Infected Hearing Impaired Infants: ValEAR Trial
Brief Title: Randomized Controlled Trial of Valganciclovir for Cytomegalovirus Infected Hearing Impaired Infants
Acronym: ValEAR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Park (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Albert Park, Chief Peds Otolaryngology, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 90760; 1U01DC014706-01A1 (NIH)
Record Dates: First submitted 2017-03-13; First posted 2017-04-11 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Cmv Congenital; CMV; Congenital Cmv; SNHL; Sensorineural Hearing Loss
Keywords: valganciclovir
MeSH Terms: conditions — Cytomegalovirus Infections; Hearing Loss, Sensorineural | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo and active drug will be dispensed in identical amber bottles with identical labeling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Valganciclovir 16 mg/kg PO twice daily (BID) x 6 months
  Interventions: Drug: Valganciclovir
- Arm B (Placebo Comparator): Flavored Simple Syrup, volume equivalent to active arm dose, PO BID x 6 months
  Interventions: Drug: Simple Syrup

INTERVENTIONS:
Drug: Valganciclovir — Valganciclovir is supplied as a powder for reconstitution into an oral solution. The reconstituted solution formulation comprises the following excipients: Povidone K30, fumaric acid, sodium benzoate, saccharin sodium, mannitol, flavor, and purified water.
  Other Names: Valcyte
  Arms: Arm A
Drug: Simple Syrup — Simple Syrup contains sucrose 85% weight by volume, purified water, and methyl paraben as a preservative along with natural preservatives. It will be flavored to match the flavor of valganciclovir.
  Other Names: Sucrose Water
  Arms: Arm B

SUMMARY:
The overall goal of this study is to determine the clinical benefit and safety of antiviral therapy for asymptomatic congenital cytomegalovirus (cCMV) infected hearing-impaired infants. We will conduct a multi-center double-blind randomized placebo-controlled trial to determine whether hearing-impaired infants with asymptomatic cCMV have better hearing and language outcomes if they receive valganciclovir antiviral treatment. We will also determine the safety of antiviral valganciclovir therapy for asymptomatic cCMV-infected hearing impaired infants. This study will be unique in that the cohort enrolled will only include hearing-impaired infants with asymptomatic cCMV.

Primary Objective: To determine if treatment of cCMV-infected hearing impaired infants with isolated hearing loss with the antiviral drug valganciclovir reduces the mean slope of total hearing thresholds over the 20 months after randomization compared to untreated cCMV-infected infants with isolated hearing loss.

Main Secondary Objectives:

1. To determine if valganciclovir treatment improves the following outcomes when compared to the control group:

   1. The slope of best ear hearing thresholds over the 20 months after randomization.
   2. The MacArthur-Bates Communicative Development Inventory (CDI) percentile score for words produced at 20 months of age.
2. To evaluate safety measures based on all grade 3 or greater new adverse events designated by the NIAID Division of AIDS (DAIDS) toxicity tables.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) can be transmitted from the mother to the fetus and is a leading cause of sensorineural hearing loss (SNHL), which is a condition where the inner ear is unable to convert sound into nerve impulses to the brain. This hearing loss and its detrimental effect on language development contribute nearly $4 billion annually to the health care costs in the U.S. Unlike other types of SNHL, CMV induced hearing loss can be treated. Several clinical trials have demonstrated that antiviral therapy may prevent progressive hearing loss if administered early in life for severely affected (symptomatic CMV) infants. These promising findings have given rise to a debate regarding the best method for identifying and treating the more numerous asymptomatic CMV-infected infants.

One approach is to conduct universal newborn hearing screens, and then do CMV diagnostic testing only on the infants who fail the hearing screen. This targeted approach should identify those infants at greatest risk of developing progressive hearing loss and consequent communicative difficulties. Utah is the first state to mandate this approach whereby infants under three weeks of age who fail their newborn hearing screening undergo CMV testing. In this trial, the hearing screen targeted approach will be used to identify patients eligible for participation in a double blind placebo controlled randomized clinical trial of antiviral valganciclovir therapy. The results of this trial will inform public policy, potentially shift our current clinical practice regarding pediatric hearing loss evaluation, and potentially offer a therapeutic option to asymptomatic CMV-infected infants with SNHL.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 1 month and less than or equal to 12 months at the time of randomization; AND
* Positive congenital CMV by urine culture or polymerase chain reaction test(PCR), OR saliva culture or PCR followed by confirmatory urine PCR by 21 days of age, OR urine culture or PCR after 21 days of age followed by newborn dry blood spot PCR; AND
* Confirmed sensorineural hearing loss (SNHL) by auditory brainstem response (ABR) testing. For ABR assessments, hearing loss is defined as levels greater than 25 dB normal hearing levels (NHL) at 1, 2, or 4 kHz in one or both ears.

Exclusion Criteria:

* Imminent demise; OR
* Known hypersensitivity reaction to valganciclovir, ganciclovir, or any components of the investigational product formulation; OR
* ALT (Alanine Aminotransferase) five times baseline U/L, hepatomegaly, or significant gastrointestinal disorders (e.g., eosinophilic esophagitis, ulcerative colitis); OR
* Absolute neutrophil count (ANC) less than 500 cells/mm^3, Hemoglobin less than 8 g/dL, or platelets less than 50,000/mm^3, splenomegaly, or significant hematologic disorders (e.g., hemophilia, leukemia, sickle cell anemia); OR
* Creatinine clearance less than 60 mL/min/1.73m^2 or significant renal disorders (e.g., nephrotic syndrome); OR
* Receiving other antiviral medications or immune globulin therapy; OR
* Receiving other investigational drugs; OR
* Breast feeding from a mother receiving antiviral or immunosuppressive medication; OR
* Known HIV positive mother (risk of immunosuppression); OR
* Subject is currently using list of prohibited medication specified by the package insert; OR
* Other known cause contributing to SNHL (e.g., meningitis, aminoglycoside ototoxicity); OR
* Bilateral profound SNHL or auditory neuropathy spectrum disorder; OR
* Existing conductive hearing loss or mixed permanent hearing loss is present; OR
* Evidence of intracranial calcification; OR
* Evidence of hydrocephalus; OR
* Microcephaly; OR
* Presence of petechiae; OR
* Intrauterine growth retardation; OR
* Chorioretinitis, optic atrophy or pale optic nerves; OR
* Parent or guardian unable to speak English or Spanish; OR
* Subject exposed to a language other than English or Spanish a majority of the time; OR
* Subject unable to complete hearing assessments or parent/guardian unable to complete communication questionnaires; OR
* < 32 weeks gestational age at birth; OR
* Weight at the time of birth < 1800 g.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Total Ear Hearing Slope | Assessed at baseline, 8, 14 and 20 months post-randomization
  The primary objective of this randomized trial is to determine if treatment of cCMV-infected infants with isolated hearing loss with the antiviral drug valganciclovir reduces the slope of the total ear hearing thresholds over the 20 months after randomization compared to that of untreated cCMV-infected infants with isolated hearing loss.

SECONDARY OUTCOMES:
Best Ear Hearing Slope | Assessed at baseline, 8, 14 and 20 months post-randomization
  The computation of the slope of the best-ear hearing thresholds begins with the same preliminary averaging steps across MRLs and truncation of threshold levels to between 15 and 110 dB as is described above for the total ear hearing slope, but in this case the analysis is based on the best-ear hearing score at each time point.
Percentile Score for Words Produced Endpoint | Assessed at 20 months of age
  The main communicative development endpoint will be determined based on the MacArthur-Bates CDI words produced percentile score given at 20 months of age.

OTHER OUTCOMES:
Words Produced Below 10th Percentile | 14 and 20 month of age assessments
  Dichotomous endpoint defined by children's communicative competency as above or below the 10th percentile based upon on the number of words produced.
Additional MacArthur Bates - Words and Sentences Subscale Percentiles | 20 month of age assessment
  The percentile scores for the MacArthur Bates Communicative Development Inventory Words and Sentences for complexity and the word form subscales, and the mean length utterance.
MacArthur Bates - Words and Gestures Subscale Percentiles | 14 months of age assessment
  Secondary communicative development endpoints will be obtained from parent report on the MacArthur Bates Communicative Development Inventory - Words and Gestures form at 14-months. The scores will be the percentile scores for the total number of words produced, total gestures, phrases understood and words understood.
Developmental Domain Endpoints | 14 and 20 months of age assessments
  Based on parent report on the Ages and Stages Questionnaire, 3rd Edition. There are five subtests on the ASQ-3. These include communication, gross motor, fine motor, problem solving, and personal- social. We will use the following scores:1)Raw scores from each subtest 2)Dichotomous endpoints for each subtest based upon the raw score above or below a designated cut-off score based upon age
Valganciclovir Pharmacokinetics | From week 2 to month 6 post-randomization
  Valganciclovir drug levels will be measured.
Viral Resistance | Assessed at month 7 post-randomization
  The presence of viral resistance will be measured.
Viral Load | Assessed at baseline month 3, and month 7 post-randomization
  Viral load will be measured
LittlEARS | 14 and 20 months of age assessments
  The raw scores will be dichotomized based on the child's hearing age and compared to standardized scores.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Park, MD, Principal Investigator — University of Utah
Locations (30):
- United States (30):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Saint Louis Universtiy, St Louis, Missouri
  - Children's Hospital at Dartmouth-Hitchcock, Lebanon, New Hampshire
  - University of New Mexico, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Weill Cornell Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cohen Children's Medical Center, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No